CLINICAL TRIAL: NCT06448936
Title: Assessment of Quality of Life in Patients Undergoing Surgery for Difficult-to-treat Basal Cell Carcinoma of the Face in Stage IIA or IIIB According to the European Association of Dermato-Oncology Classification.
Brief Title: Quality of Life in Patients With Difficult-to-Treat Basal Cell Carcinoma: An Evaluation of Impact and Surgical Outcomes.
Acronym: FACE-QOL
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6722
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-05

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient-reported outcome measures (PROMs) — Administration of questionnaires investigating the impact of facial difficult-to-treat basal cell carcinoma treated by surgery on patient's quality of life over the course of one year. The questionnaires will be submitted at baseline (i.e., before surgery) and at 3-months follow up.
  Other Names: GHQ-12 Questionnaire; Skindex-17 Questionnaire; PRISM Questionnaire; NAFEQ Questionnaire; Skin Cancer Index Questionnaire

SUMMARY:
FACE-QoL is an observational, prospective, multicenter study aimed at evaluating the impact of surgical treatment on quality of life in patients with stage IIA and IIIB difficult-to-treat basal cell carcinoma of the face, according to the European Academy of Dermato-Oncology classification, using patient-reported outcomes.

The main questions the study seeks to answer are:

Can surgery, as the gold standard treatment, lead to an improvement in the quality of life of patients with difficult-to-treat basal cell carcinoma in functionally and cosmetically challenging sites of the face (i.e., stage IIA and IIIB)? Which clinical and individual variables have the greatest impact on patients' quality of life? Participants will complete questionnaires assessing their quality of life and the impact of the disease on their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or histological diagnosis of difficult-to-treat basal cell carcinoma (DTT-BCC) classified as stage IIA or IIIB according to the EADO classification.
* Tumor location: face.
* Intervention: surgical treatment of facial stage IIA and IIIB difficult-to-treat basal cell carcinoma.
* Sufficient knowledge of spoken and written Italian by the patient.

Exclusion Criteria:

* Known psychiatric or substance abuse disorders that may interfere with cooperation and compliance with trial requirements.
* Inoperable or metastatic difficult-to-treat basal cell carcinoma.
* Contraindications to surgery related to the patient's condition.
* Previous radiation therapy involving the field of the target lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sequential recruitment of patients undergoing surgery for difficult-to-treat basal cell carcinoma of the face in stage IIA or IIIB, according to the European Association of Dermato-Oncology (EADO) classification.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Surgery in difficult-to-treat basal cell carcinoma | 1 year
  The primary outcome is to assess the change in quality of life in patients with difficult-to-treat basal cell carcinoma (DTT-BCC) of the face (stage IIA and IIIB according to the European Association of Dermato-Oncology classification) before and after surgery, as measured by various questionnaires.

SECONDARY OUTCOMES:
Predictive variables | 1 year
  A secondary endpoint is to identify which clinical and individual variables have the greatest impact on patients' quality of life (e.g., age, gender, tumor site or size, primary vs. recurrent, type of reconstruction, etc.).
Validation of the NAFEQ score. | 1 year
  A secondary endpoint is to validate the Italian version of the NAFEQ score (Nasal Appearance and Function Evaluation Questionnaire) to assess the impact of surgery on quality of life in patients with DTT-BCCs of the nose (including various nasal subunits, such as the dorsum, ala, side wall, tip, etc.). The questionnaire consists of 14 questions directed to patients, with a total score ranging from 18 to 66, where a score of 66 indicates post-surgical clinical and aesthetic improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Paradisi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy